CLINICAL TRIAL: NCT04830059
Title: The Joint Effect of Air Pollution and Exercise on Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tsinghua University (Other)
Responsible Party: Principal Investigator, Jianxiu Liu, Research staff, Tsinghua University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: THU2021
Record Dates: First submitted 2021-03-29; First posted 2021-04-02 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2021-04

CONDITIONS: Exercise; Air Pollution; Cognition; Health Promotion
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Double blind randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and investigators are blinded, and part of the outcome assessors are blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- High intensity intermittent training (Experimental): HIIT exercise program: 20 minutes HIIT exercise (1min 100% VO2max and 1min 50% VO2max alternately), and warm-up and relaxation before and after exercise for 10 minutes.
  Interventions: Behavioral: Exercise
- HIIT with pollution reduction (Experimental): HIIT program: 20 minutes HIIT exercise (1min 100% VO2max and 1min 50% VO2max alternately), and warm-up and relaxation before and after exercise for 10 minutes; Environmental pollution intervention program: air purification system is used order to reduce the PM2.5 and PM10.
  Interventions: Behavioral: Exercise; Behavioral: Air purification
- Moderate intensity continuous training (Experimental): MICT program: 20 minutes of 70-75% VO2max exercise and 10 minutes of warm-up and relaxation before and after exercise.
  Interventions: Behavioral: Exercise
- MICT with pollution reduction (Experimental): MICT program: 20 minutes of 70-75% VO2max exercise and 10 minutes of warm-up and relaxation before and after exercise; Environmental pollution intervention program: air purification system is used order to reduce the PM2.5 and PM10.
  Interventions: Behavioral: Exercise; Behavioral: Air purification
- Stretch control group (Experimental): Stretching control group: 30 minutes stretching, posture adjustment and rehabilitation courses is taught by professional therapist.
  Interventions: Behavioral: Exercise
- Control with pollution reduction (Experimental): Stretching control group: 30 minutes stretching, posture adjustment and rehabilitation courses is taught by professional therapist.
  Environmental pollution intervention program: air purification system is used order to reduce the PM2.5 and PM10.
  Interventions: Behavioral: Exercise; Behavioral: Air purification

INTERVENTIONS:
Behavioral: Exercise — Two types of exercise intervention and control group
Behavioral: Air purification — Air purification in order to reduce the PM2.5 and PM10
  Arms: Control with pollution reduction; HIIT with pollution reduction; MICT with pollution reduction

SUMMARY:
A double-blind randomized controlled trial design is used in this study. A mixed design of 2 (pollution reduction group vs. no pollution reduction group) × 3 (high intensity intermittent exercise [HIIT], moderate intensity of aerobic exercise [MICT] and control group [CONT]) is used. 93 subjects recruited by advertising will be randomly divided into 6 groups: high intensity exercise group (pollution reduction vs no pollution reduction), moderate intensity aerobic exercise group (pollution reduction vs no pollution reduction) and Stretching group (Control) (pollution reduction vs no pollution reduction).

DETAILED DESCRIPTION:
Environmental intervention program In the pollution reduction groups, the air purification system is used 2 hours before the subjects entered the room to minimize the indoor PM2.5 and PM10.

Exercise intervention program including HIIT, MICT and Stretching (Control) group :

The VO2max of all subjects are measured one week before the experiment. HIIT program: 20 minutes exercise of HIIT (1min of 100% VO2max and 1min of 50% VO2max alternately) and 10 minutes of warm-up and relaxation.

MICT program: 20 minutes exercise of 70-75% VO2max and 10 minutes of warm-up and relaxation.

Stretching control group: 30 minutes of stretching, posture adjustment and rehabilitation courses taught by professional therapists.

ELIGIBILITY:
Inclusion Criteria:

* No regular exercise in the past six months;
* Healthy people without history of disease;
* Aged between 20 and 30 years old.

Exclusion Criteria:

* Professional athletes;
* Regular exercise in the past six months;
* People who are injured or have a history of disease in the past six months;
* People who have a history of taking medicine in the past six months.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Change of cognitive function | Before and after acute exercise (about 30 minutes).
  Cognitive function measured by computer-based tasks including executive function
Change of biomarkers | Before and after acute exercise (about 30 minutes).
  The cognitive-related biomarkers including brain derived neurotrophic factor
Change of oxyhemoglobin | Before and after acute exercise (about 30 minutes).
  Mearsurement of oxyhemoglobin using fNIRS
Change of transcriptions | Before and after acute exercise (about 30 minutes).
  The molecular response of exercise and environment through the measurement of peripheral blood
Change of metabonomics | Before and after acute exercise (about 30 minutes).
  The molecular response of exercise and environment through the measurement of peripheral blood
Change of cerebral blood flow | Before and after acute exercise (about 30 minutes).
  The blood flow of middle cerebral artery measured by ultrasonic doppler

SECONDARY OUTCOMES:
Change of cognitive function | Three months (from baseline to the third month)
  Cognitive function measured by computer-based tasks including executive function
Change of aerobic capacity | Three months (from baseline to the third month)
  The aerobic capacity measured by the gas metabolism analyzer
Change of cerebral blood flow | Three months (from baseline to the third month)
  The blood flow of middle cerebral artery measured by ultrasonic doppler
Change of biomarkers | Three months (from baseline to the third month)
  The cognitive-related biomarkers including brain derived neurotrophic factor
Change of oxyhemoglobin | Three months (from baseline to the third month)
  Mearsurement of oxyhemoglobin using functional near infrared spectroscopy
Change of metabonomics | Three months (from baseline to the third month)
  The molecular response of exercise through the measurement of peripheral blood
Change of transcriptions | Three months (from baseline to the third month)
  The molecular response of exercise through the measurement of peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Qian Di, Sc.D., Study Director — Wanke School of public health, Tsinghua University; Xindong Ma, PhD, Study Chair — Department of physical education, Tsinghua University
Locations (1):
- Tsinghua University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Liu J, Min L, Liu R, Zhang X, Wu M, Di Q, Ma X. The effect of exercise on cerebral blood flow and executive function among young adults: a double-blinded randomized controlled trial. Sci Rep. 2023 May 22;13(1):8269. doi: 10.1038/s41598-023-33063-9. PMID 37217511
- [Derived] Liu J, Zhang Y, Li X, Wang D, Shi B, You Y, Min L, Luo B, Li Y, Di Q, Ma X. Exercise improves mental health status of young adults via attenuating inflammation factors but modalities matter. Front Psychiatry. 2022 Dec 14;13:1067890. doi: 10.3389/fpsyt.2022.1067890. eCollection 2022. PMID 36590621